CLINICAL TRIAL: NCT04650386
Title: Enhancing Office-based Buprenorphine Treatment: An Adaptive Psychosocial Approach
Brief Title: Examining an Adaptive Approach to Providing Psychosocial Support to Buprenorphine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Management Corporation (Other)
Collaborators: Philadelphia College of Osteopathic Medicine (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1908
Record Dates: First submitted 2020-11-05; First posted 2020-12-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Opioid-use Disorder
Keywords: Opioid Use; Medication Assisted Treatment; Psychosocial Treatment; Cognitive Behavioral Therapy; Peer Support; Peer Recovery Specialist; Certified Recovery Specialist; Opioid Use Disorder; Adaptive Intervention; Office-Based Opioid Treatment; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): Participants assigned to the TAU condition will be scheduled for buprenorphine medication management appointments and will receive OBOT at the FQHC and adjunctive psychosocial treatment as typically provided at the FQHC. The team will continue to meet with the patient during subsequent MAT visits on a decreasing frequency, with some slight site-specific variation. The schedule of MAT visits generally includes 3 clinic visits during the week of induction, 1-2 visits per week until the patient is stabilized, and monthly thereafter. Behavioral health clinicians provide support to the patient, discuss UDS results, assist with strategic problem-solving around recovery and adjustment to sobriety, and monitor the patient's engagement in MAT.
- Adaptive Intervention (Experimental): Participants assigned to the adaptive intervention condition will be scheduled for buprenorphine medication management appointments according to the clinic protocol described above for TAU. The adjunctive psychosocial treatment that participants in this condition receive are (1) CBT delivered by behavioral health specialists and/or (2) peer support delivered by certified recovery specialist. The active intervention period will span 3 months post-study entry. Participants will continue to receive TAU following the active intervention period.
  Interventions: Behavioral: Psychosocial support determined by adaptive treatment algorithm

INTERVENTIONS:
Behavioral: Psychosocial support determined by adaptive treatment algorithm — Participants assigned to the adaptive intervention condition will be scheduled for buprenorphine medication management appointments according to the clinic protocol described above for TAU. The adjunctive psychosocial treatment that participants in this condition receive are (1) CBT delivered by behavioral health specialists and/or (2) peer support delivered by certified recovery specialist. The active intervention period will span 3 months post-study entry. Participants will continue to receive TAU following the active intervention period.
  Arms: Adaptive Intervention

SUMMARY:
The purpose of this study is to address important knowledge gaps regarding the optimal way to provide psychosocial treatment to patients who are receiving buprenorphine for opioid use disorder (OUD) in office-based settings. The project will develop and evaluate an adaptive treatment approach in which the interventions are delivered based on the individual needs of patients at baseline and throughout the course of care. The adaptive intervention will incorporate certified recovery specialists (CRSs) and cognitive behavioral therapy (CBT), two interventions that have been widely used in the treatment of OUD. The efficacy of the adaptive intervention will be evaluated through a randomized controlled trial (RCT) that will be conducted in federally qualified health (FQHCs) in Philadelphia.

DETAILED DESCRIPTION:
This study will help to inform best practices for providing psychosocial treatment within the context of office-based opioid treatment (OBOT) with buprenorphine. We will use a staged approach to develop and evaluate an adaptive approach to the provision of adjunctive psychosocial treatment that includes medication management by a buprenorphine provider and linkage to CRSs and CBT depending on the needs of the patient. The specific aims of the proposal are listed below.

Aim 1: Work collaboratively with our multidisciplinary team to develop specific protocols for the CRS and CBT interventions and establish algorithms based on behavioral criteria to determine when each intervention should be implemented. As a part of this aim, we will also develop standard procedures for delivering each intervention and train interventionists [i.e., CRSs and Licensed Professional Counselors (LPCs)] to deliver them with fidelity.

Aim 2: Conduct a two-group randomized study to evaluate the efficacy of the adaptive intervention relative to TAU. Outcomes to be examined will include urinalysis-confirmed opioid use, retention in buprenorphine- based OBOT, quality of life, and psychosocial functioning through one year post-study entry.

Aim 3: Conduct a qualitative evaluation of the intervention and develop a strategic plan for its dissemination. We will conduct focus groups with clinic staff and relevant stakeholders to determine the utility and acceptability of the adaptive intervention. In addition, we will hold an expert roundtable to identify mechanisms for increasing sustainability and enhancing adoption by other office-based buprenorphine programs to inform the development of the strategic plan.

Aim 4: Establish a training program in clinical research for minority students. Eight undergraduate students from a historically minority higher education institution will be selected to participate in 9-month internships during which they will receive comprehensive and pragmatic training in the full range of clinical research from study design to dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Have initiated office-based buprenorphine treatment for OUD at the FQHC within the last 4 weeks;
* Not require an inpatient level of care as determined by the healthcare provider; and
* Be capable of providing valid contact information and informed consent.

Exclusion Criteria:

* Patient is under the age of 18;
* Co-morbid psychiatric disorder indicating the need for more intensive residential treatment
* Patient is unable to provide informed consent.

Individuals who are intoxicated, cognitively impaired, or psychiatrically unstable at baseline will not be included; however, they may subsequently be included if the disqualifying condition subsides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Urinalysis-confirmed abstinence from opioids at 3 month follow up | 3 months post study entry
  Participants will provide a urine specimen at the 3 month follow up assessment. We will use the CLIA Waived® 14-Panel Drug Test Cup and fentanyl test strip for opioids, buprenorphine, methadone, oxycodone, THC, cocaine, amphetamines, PCP, methamphetamine, benzodiazepines, and barbiturates, and MDMD. The urine sample will be delivered under the supervision of the RA who will use standard procedures to detect tampering and dilution.
Urinalysis-confirmed abstinence from opioids at 6 month follow up | 6 months post study entry
  Participants will provide a urine specimen at the 6 month follow up assessment. We will use the CLIA Waived® 14-Panel Drug Test Cup and fentanyl test strip for opioids, buprenorphine, methadone, oxycodone, THC, cocaine, amphetamines, PCP, methamphetamine, benzodiazepines, and barbiturates, and MDMD. The urine sample will be delivered under the supervision of the RA who will use standard procedures to detect tampering and dilution.
Urinalysis-confirmed abstinence from opioids at 9 month follow up | 9 months post study entry
  Participants will provide a urine specimen at the 9 month follow up assessment. We will use the CLIA Waived® 14-Panel Drug Test Cup and fentanyl test strip for opioids, buprenorphine, methadone, oxycodone, THC, cocaine, amphetamines, PCP, methamphetamine, benzodiazepines, and barbiturates, and MDMD. The urine sample will be delivered under the supervision of the RA who will use standard procedures to detect tampering and dilution.
Urinalysis-confirmed abstinence from opioids at 12 month follow up | 12 months post study entry
  Participants will provide a urine specimen at the 12 month follow up assessment. We will use the CLIA Waived® 14-Panel Drug Test Cup and fentanyl test strip for opioids, buprenorphine, methadone, oxycodone, THC, cocaine, amphetamines, PCP, methamphetamine, benzodiazepines, and barbiturates, and MDMD. The urine sample will be delivered under the supervision of the RA who will use standard procedures to detect tampering and dilution.

SECONDARY OUTCOMES:
Abstinence from or reductions in use of other (non-opioid) psychoactive substances | Through 12 months post-study entry
  Results from the CLIAwaived® 14-panel test and fentanyl strip described above for the primary outcome will be used as an indicator of this outcome.
Retention in buprenorphine-based OBOT | Through 12 months post-study entry
  Including appointment attendance, medication and treatment adherence, and retention in and completion of treatment.
Quality of life assessment | Through 12 months post-study entry
  Quality of life will be measured using the Short Form-36 (SF-36). The SF-36 is a self-report inventory that assesses eight dimensions of physical and mental health-related quality of life. The SF-36 has been shown to have high reliability and validity.
Psychosocial functioning/Multidimensional problem severity | Through 12 months post-study entry
  Multidimensional problem severity, a secondary outcome, will be measured using the Addiction Severity Index-Lite (ASI-Lite). The ASI-Lite is a reliable and valid multidimensional assessment that provides composite scores reflecting current problem severity in the medical, employment, alcohol, drug, legal, family/social, and psychiatric areas.
Treatment satisfaction | Through 12 months post-study entry
  Treatment satisfaction will be measured using a modified version of the Treatment Services Review (TSR). The TSR measures patient therapeutic engagement in and satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Dugosh, Ph.D., Principal Investigator — PHMC
Locations (2):
- United States (2):
  - Project HOME Stephen J. Klein Wellness Center, Philadelphia, Pennsylvania
  - PHMC Care Clinic, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato L, Minozzi S, Davoli M, Vecchi S. Psychosocial and pharmacological treatments versus pharmacological treatments for opioid detoxification. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD005031. doi: 10.1002/14651858.CD005031.pub4. PMID 21901695
- [Background] Alford DP, LaBelle CT, Kretsch N, Bergeron A, Winter M, Botticelli M, Samet JH. Collaborative care of opioid-addicted patients in primary care using buprenorphine: five-year experience. Arch Intern Med. 2011 Mar 14;171(5):425-31. doi: 10.1001/archinternmed.2010.541. PMID 21403039
- [Background] Andraka-Christou B, Capone MJ. A qualitative study comparing physician-reported barriers to treating addiction using buprenorphine and extended-release naltrexone in U.S. office-based practices. Int J Drug Policy. 2018 Apr;54:9-17. doi: 10.1016/j.drugpo.2017.11.021. Epub 2018 Jan 8. PMID 29324253
- [Background] Araya R, Rojas G, Fritsch R, Gaete J, Rojas M, Simon G, Peters TJ. Treating depression in primary care in low-income women in Santiago, Chile: a randomised controlled trial. Lancet. 2003 Mar 22;361(9362):995-1000. doi: 10.1016/S0140-6736(03)12825-5. PMID 12660056
- [Background] Barry DT, Irwin KS, Jones ES, Becker WC, Tetrault JM, Sullivan LE, Hansen H, O'Connor PG, Schottenfeld RS, Fiellin DA. Integrating buprenorphine treatment into office-based practice: a qualitative study. J Gen Intern Med. 2009 Feb;24(2):218-25. doi: 10.1007/s11606-008-0881-9. Epub 2008 Dec 17. PMID 19089500
- [Background] Bassuk EL, Hanson J, Greene RN, Richard M, Laudet A. Peer-Delivered Recovery Support Services for Addictions in the United States: A Systematic Review. J Subst Abuse Treat. 2016 Apr;63:1-9. doi: 10.1016/j.jsat.2016.01.003. Epub 2016 Jan 13. PMID 26882891
- [Background] Beck AT. Cognitive therapy : nature and relation to behavior therapy. J Psychother Pract Res. 1993 Fall;2(4):342-56. No abstract available. PMID 22700159
- [Background] Breslin FC, Sobell MB, Sobell LC, Cunningham JA, Sdao-Jarvie K, Borsoi D. Problem drinkers: evaluation of a stepped-care approach. J Subst Abuse. 1998;10(3):217-32. doi: 10.1016/s0899-3289(99)00008-5. PMID 10689656
- [Background] Brooner RK, Kidorf M. Using behavioral reinforcement to improve methadone treatment participation. Sci Pract Perspect. 2002 Jul;1(1):38-47. doi: 10.1151/spp021138. PMID 18567965
- [Background] Brooner RK, Kidorf MS, King VL, Stoller KB, Peirce JM, Bigelow GE, Kolodner K. Behavioral contingencies improve counseling attendance in an adaptive treatment model. J Subst Abuse Treat. 2004 Oct;27(3):223-32. doi: 10.1016/j.jsat.2004.07.005. PMID 15501375
- [Background] Brooner RK, Kidorf MS, King VL, Stoller KB, Neufeld KJ, Kolodner K. Comparing adaptive stepped care and monetary-based voucher interventions for opioid dependence. Drug Alcohol Depend. 2007 May;88 Suppl 2(Suppl 2):S14-23. doi: 10.1016/j.drugalcdep.2006.12.006. Epub 2007 Jan 24. PMID 17257782
- [Background] Cacciola JS, Alterman AI, McLellan AT, Lin YT, Lynch KG. Initial evidence for the reliability and validity of a "Lite" version of the Addiction Severity Index. Drug Alcohol Depend. 2007 Mar 16;87(2-3):297-302. doi: 10.1016/j.drugalcdep.2006.09.002. Epub 2006 Oct 11. PMID 17045423
- [Background] Carels RA, Darby L, Cacciapaglia HM, Douglass OM, Harper J, Kaplar ME, Konrad K, Rydin S, Tonkin K. Applying a stepped-care approach to the treatment of obesity. J Psychosom Res. 2005 Dec;59(6):375-83. doi: 10.1016/j.jpsychores.2005.06.060. PMID 16310019
- [Background] Choi NG, DiNitto DM, Marti CN. Treatment use, perceived need, and barriers to seeking treatment for substance abuse and mental health problems among older adults compared to younger adults. Drug Alcohol Depend. 2014 Dec 1;145:113-20. doi: 10.1016/j.drugalcdep.2014.10.004. Epub 2014 Oct 16. PMID 25456572
- [Background] Collins LM, Murphy SA, Bierman KL. A conceptual framework for adaptive preventive interventions. Prev Sci. 2004 Sep;5(3):185-96. doi: 10.1023/b:prev.0000037641.26017.00. PMID 15470938
- [Background] Dugosh K, Abraham A, Seymour B, McLoyd K, Chalk M, Festinger D. A Systematic Review on the Use of Psychosocial Interventions in Conjunction With Medications for the Treatment of Opioid Addiction. J Addict Med. 2016 Mar-Apr;10(2):93-103. doi: 10.1097/ADM.0000000000000193. PMID 26808307
- [Background] Dugosh KL, Festinger DS, Croft JR, Marlowe DB. Measuring coercion to participate in research within a doubly vulnerable population: initial development of the coercion assessment scale. J Empir Res Hum Res Ethics. 2010 Mar;5(1):93-102. doi: 10.1525/jer.2010.5.1.93. PMID 20235867
- [Background] Dutra L, Stathopoulou G, Basden SL, Leyro TM, Powers MB, Otto MW. A meta-analytic review of psychosocial interventions for substance use disorders. Am J Psychiatry. 2008 Feb;165(2):179-87. doi: 10.1176/appi.ajp.2007.06111851. Epub 2008 Jan 15. PMID 18198270
- [Background] Dryden W, Bond FW. Reason and emotion in psychotherapy: Albert Ellis. Br J Psychiatry. 1994 Jul;165(1):131-5. doi: 10.1192/bjp.165.1.131. PMID 7953024
- [Background] Festinger DS, Marlowe DB, Lee PA, Kirby KC, Bovasso G, McLellan AT. Status hearings in drug court: when more is less and less is more. Drug Alcohol Depend. 2002 Oct 1;68(2):151-7. doi: 10.1016/s0376-8716(02)00187-4. PMID 12234644
- [Background] Fiellin DA, Barry DT, Sullivan LE, Cutter CJ, Moore BA, O'Connor PG, Schottenfeld RS. A randomized trial of cognitive behavioral therapy in primary care-based buprenorphine. Am J Med. 2013 Jan;126(1):74.e11-7. doi: 10.1016/j.amjmed.2012.07.005. PMID 23260506
- [Background] Fiellin DA, Moore BA, Sullivan LE, Becker WC, Pantalon MV, Chawarski MC, Barry DT, O'Connor PG, Schottenfeld RS. Long-term treatment with buprenorphine/naloxone in primary care: results at 2-5 years. Am J Addict. 2008 Mar-Apr;17(2):116-20. doi: 10.1080/10550490701860971. PMID 18393054
- [Background] Fox AD, Sohler NL, Starrels JL, Ning Y, Giovanniello A, Cunningham CO. Pain is not associated with worse office-based buprenorphine treatment outcomes. Subst Abus. 2012;33(4):361-5. doi: 10.1080/08897077.2011.638734. PMID 22989279
- [Background] Haddad MS, Zelenev A, Altice FL. Integrating buprenorphine maintenance therapy into federally qualified health centers: real-world substance abuse treatment outcomes. Drug Alcohol Depend. 2013 Jul 1;131(1-2):127-35. doi: 10.1016/j.drugalcdep.2012.12.008. Epub 2013 Jan 17. PMID 23332439
- [Background] Inocencio TJ, Carroll NV, Read EJ, Holdford DA. The economic burden of opioid-related poisoning in the United States. Pain Med. 2013 Oct;14(10):1534-47. doi: 10.1111/pme.12183. Epub 2013 Jul 10. PMID 23841538
- [Background] Jenkinson C, Layte R, Jenkinson D, Lawrence K, Petersen S, Paice C, Stradling J. A shorter form health survey: can the SF-12 replicate results from the SF-36 in longitudinal studies? J Public Health Med. 1997 Jun;19(2):179-86. doi: 10.1093/oxfordjournals.pubmed.a024606. PMID 9243433
- [Background] Kampman K, Jarvis M. American Society of Addiction Medicine (ASAM) National Practice Guideline for the Use of Medications in the Treatment of Addiction Involving Opioid Use. J Addict Med. 2015 Sep-Oct;9(5):358-67. doi: 10.1097/ADM.0000000000000166. PMID 26406300
- [Background] Kidorf M, Neufeld K, Brooner RK. Combining stepped-care approaches with behavioral reinforcement to motivate employment in opioid-dependent outpatients. Subst Use Misuse. 2004;39(13-14):2215-38. doi: 10.1081/ja-200034591. PMID 15603002
- [Background] Kidorf M, Neufeld K, King VL, Clark M, Brooner RK. A stepped care approach for reducing cannabis use in opioid-dependent outpatients. J Subst Abuse Treat. 2007 Jun;32(4):341-7. doi: 10.1016/j.jsat.2006.09.005. Epub 2006 Dec 11. PMID 17481457
- [Background] King VL, Stoller KB, Hayes M, Umbricht A, Currens M, Kidorf MS, Carter JA, Schwartz R, Brooner RK. A multicenter randomized evaluation of methadone medical maintenance. Drug Alcohol Depend. 2002 Jan 1;65(2):137-48. doi: 10.1016/s0376-8716(01)00155-7. PMID 11772475
- [Background] Kissin W, McLeod C, Sonnefeld J, Stanton A. Experiences of a national sample of qualified addiction specialists who have and have not prescribed buprenorphine for opioid dependence. J Addict Dis. 2006;25(4):91-103. doi: 10.1300/J069v25n04_09. PMID 17088229
- [Background] Kumari S, Manalai P, Leong S, Wooditch A, Malik M, Lawson WB. Factors associated with non-adherence to Buprenorphine-naloxone among opioid dependent African-Americans: A retrospective chart review. Am J Addict. 2016 Mar;25(2):110-7. doi: 10.1111/ajad.12325. Epub 2016 Jan 8. PMID 26749158
- [Background] Lavori PW. Clinical trials in psychiatry: should protocol deviation censor patient data? Neuropsychopharmacology. 1992 Jan;6(1):39-48; discussion 49-63. PMID 1571068
- [Background] Lee CS, Liebschutz JM, Anderson BJ, Stein MD. Hospitalized opioid-dependent patients: Exploring predictors of buprenorphine treatment entry and retention after discharge. Am J Addict. 2017 Oct;26(7):667-672. doi: 10.1111/ajad.12533. Epub 2017 Mar 21. PMID 28324627
- [Background] Lee JD, Nunes EV Jr, Novo P, Bachrach K, Bailey GL, Bhatt S, Farkas S, Fishman M, Gauthier P, Hodgkins CC, King J, Lindblad R, Liu D, Matthews AG, May J, Peavy KM, Ross S, Salazar D, Schkolnik P, Shmueli-Blumberg D, Stablein D, Subramaniam G, Rotrosen J. Comparative effectiveness of extended-release naltrexone versus buprenorphine-naloxone for opioid relapse prevention (X:BOT): a multicentre, open-label, randomised controlled trial. Lancet. 2018 Jan 27;391(10118):309-318. doi: 10.1016/S0140-6736(17)32812-X. Epub 2017 Nov 14. PMID 29150198
- [Background] Ling W, Hillhouse M, Ang A, Jenkins J, Fahey J. Comparison of behavioral treatment conditions in buprenorphine maintenance. Addiction. 2013 Oct;108(10):1788-98. doi: 10.1111/add.12266. Epub 2013 Jul 12. PMID 23734858
- [Background] Litz M, Leslie D. The impact of mental health comorbidities on adherence to buprenorphine: A claims based analysis. Am J Addict. 2017 Dec;26(8):859-863. doi: 10.1111/ajad.12644. Epub 2017 Nov 16. PMID 29143483
- [Background] Marlowe DB, Festinger DS, Dugosh KL, Arabia PL, Kirby KC. An effectiveness trial of contingency management in a felony preadjudication drug court. J Appl Behav Anal. 2008 Winter;41(4):565-77. doi: 10.1901/jaba.2008.41-565. PMID 19192860
- [Background] Marlowe DB, Festinger DS, Dugosh KL, Benasutti KM, Fox G, Croft JR. Adaptive Programming Improves Outcomes in Drug Court: An Experimental Trial. Crim Justice Behav. 2012 Apr 1;39(4):514-532. doi: 10.1177/0093854811432525. PMID 22923854
- [Background] Marlowe DB, Festinger DS, Dugosh KL, Benasutti KM, Fox G, Harron A. An Experimental Trial of Adaptive Programming in Drug Court: Outcomes at 6, 12 and 18 Months. J Exp Criminol. 2014 Jun 1;10(2):129-149. doi: 10.1007/s11292-013-9196-x. PMID 25346652
- [Background] Marlowe DB, Festinger DS, Dugosh KL, Lee PA, Benasutti KM. Adapting judicial supervision to the risk level of drug offenders: discharge and 6-month outcomes from a prospective matching study. Drug Alcohol Depend. 2007 May;88 Suppl 2(Suppl 2):S4-13. doi: 10.1016/j.drugalcdep.2006.10.001. Epub 2006 Oct 30. PMID 17071020
- [Background] Guidelines for the Psychosocially Assisted Pharmacological Treatment of Opioid Dependence. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK143185/ PMID 23762965
- [Background] Weiss RD, Potter JS, Fiellin DA, Byrne M, Connery HS, Dickinson W, Gardin J, Griffin ML, Gourevitch MN, Haller DL, Hasson AL, Huang Z, Jacobs P, Kosinski AS, Lindblad R, McCance-Katz EF, Provost SE, Selzer J, Somoza EC, Sonne SC, Ling W. Adjunctive counseling during brief and extended buprenorphine-naloxone treatment for prescription opioid dependence: a 2-phase randomized controlled trial. Arch Gen Psychiatry. 2011 Dec;68(12):1238-46. doi: 10.1001/archgenpsychiatry.2011.121. Epub 2011 Nov 7. PMID 22065255
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Vogt DS, King DW, King LA. Focus groups in psychological assessment: enhancing content validity by consulting members of the target population. Psychol Assess. 2004 Sep;16(3):231-43. doi: 10.1037/1040-3590.16.3.231. PMID 15456379
- [Background] Tesema L, Marshall J, Hathaway R, Pham C, Clarke C, Bergeron G, Yeh J, Soliman M, McCormick D. Training in office-based opioid treatment with buprenorphine in US residency programs: A national survey of residency program directors. Subst Abus. 2018;39(4):434-440. doi: 10.1080/08897077.2018.1449047. Epub 2018 May 14. PMID 29513136
- [Background] Center for Substance Abuse Treatment. Clinical Guidelines for the Use of Buprenorphine in the Treatment of Opioid Addiction. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2004. Report No.: (SMA) 04-3939. Available from http://www.ncbi.nlm.nih.gov/books/NBK64245/ PMID 22514846
- [Background] Stein BD, Dick AW, Sorbero M, Gordon AJ, Burns RM, Leslie DL, Pacula RL. A population-based examination of trends and disparities in medication treatment for opioid use disorders among Medicaid enrollees. Subst Abus. 2018;39(4):419-425. doi: 10.1080/08897077.2018.1449166. Epub 2018 Jun 22. PMID 29932847
- [Background] Sobell MB, Sobell LC. Stepped care as a heuristic approach to the treatment of alcohol problems. J Consult Clin Psychol. 2000 Aug;68(4):573-9. PMID 10965632
- [Background] Reif S, Braude L, Lyman DR, Dougherty RH, Daniels AS, Ghose SS, Salim O, Delphin-Rittmon ME. Peer recovery support for individuals with substance use disorders: assessing the evidence. Psychiatr Serv. 2014 Jul;65(7):853-61. doi: 10.1176/appi.ps.201400047. PMID 24838535
- [Background] Paulozzi LJ, Kilbourne EM, Desai HA. Prescription drug monitoring programs and death rates from drug overdose. Pain Med. 2011 May;12(5):747-54. doi: 10.1111/j.1526-4637.2011.01062.x. Epub 2011 Feb 18. PMID 21332934
- [Background] O'Malley SS, Rounsaville BJ, Farren C, Namkoong K, Wu R, Robinson J, O'Connor PG. Initial and maintenance naltrexone treatment for alcohol dependence using primary care vs specialty care: a nested sequence of 3 randomized trials. Arch Intern Med. 2003 Jul 28;163(14):1695-704. doi: 10.1001/archinte.163.14.1695. PMID 12885685
- [Background] Netherland J, Botsko M, Egan JE, Saxon AJ, Cunningham CO, Finkelstein R, Gourevitch MN, Renner JA, Sohler N, Sullivan LE, Weiss L, Fiellin DA; BHIVES Collaborative. Factors affecting willingness to provide buprenorphine treatment. J Subst Abuse Treat. 2009 Apr;36(3):244-51. doi: 10.1016/j.jsat.2008.06.006. Epub 2008 Aug 20. PMID 18715741
- [Background] Murphy SA, Lynch KG, Oslin D, McKay JR, TenHave T. Developing adaptive treatment strategies in substance abuse research. Drug Alcohol Depend. 2007 May;88 Suppl 2(Suppl 2):S24-30. doi: 10.1016/j.drugalcdep.2006.09.008. Epub 2006 Oct 23. PMID 17056207
- [Background] Murphy SA. An experimental design for the development of adaptive treatment strategies. Stat Med. 2005 May 30;24(10):1455-81. doi: 10.1002/sim.2022. PMID 15586395
- [Background] Morgan K, Lee J, Sebar B. Community health workers: a bridge to healthcare for people who inject drugs. Int J Drug Policy. 2015 Apr;26(4):380-7. doi: 10.1016/j.drugpo.2014.11.001. Epub 2014 Nov 13. PMID 25477284
- [Background] Moore BA, Fiellin DA, Barry DT, Sullivan LE, Chawarski MC, O'Connor PG, Schottenfeld RS. Primary care office-based buprenorphine treatment: comparison of heroin and prescription opioid dependent patients. J Gen Intern Med. 2007 Apr;22(4):527-30. doi: 10.1007/s11606-007-0129-0. PMID 17372805
- [Background] Moore BA, Barry DT, Sullivan LE, O'connor PG, Cutter CJ, Schottenfeld RS, Fiellin DA. Counseling and directly observed medication for primary care buprenorphine maintenance: a pilot study. J Addict Med. 2012 Sep;6(3):205-11. doi: 10.1097/ADM.0b013e3182596492. PMID 22614936
- [Background] McLellan AT, Cacciola JC, Alterman AI, Rikoon SH, Carise D. The Addiction Severity Index at 25: origins, contributions and transitions. Am J Addict. 2006 Mar-Apr;15(2):113-24. doi: 10.1080/10550490500528316. PMID 16595348
- [Background] McKay JR, Van Horn DH, Lynch KG, Ivey M, Cary MS, Drapkin ML, Coviello DM, Plebani JG. An adaptive approach for identifying cocaine dependent patients who benefit from extended continuing care. J Consult Clin Psychol. 2013 Dec;81(6):1063-73. doi: 10.1037/a0034265. Epub 2013 Sep 16. PMID 24041231
- [Background] McKay JR, Lynch KG, Shepard DS, Pettinati HM. The effectiveness of telephone-based continuing care for alcohol and cocaine dependence: 24-month outcomes. Arch Gen Psychiatry. 2005 Feb;62(2):199-207. doi: 10.1001/archpsyc.62.2.199. PMID 15699297
- [Background] McKay JR, Drapkin ML, Van Horn DH, Lynch KG, Oslin DW, DePhilippis D, Ivey M, Cacciola JS. Effect of patient choice in an adaptive sequential randomization trial of treatment for alcohol and cocaine dependence. J Consult Clin Psychol. 2015 Dec;83(6):1021-32. doi: 10.1037/a0039534. Epub 2015 Jul 27. PMID 26214544
- [Background] McHugh RK, Hearon BA, Otto MW. Cognitive behavioral therapy for substance use disorders. Psychiatr Clin North Am. 2010 Sep;33(3):511-25. doi: 10.1016/j.psc.2010.04.012. PMID 20599130
- [Background] Matejkowski, J., Dugosh, K. L., Clements, N. T., & Festinger, D. S. (2015). Pilot Testing of an Online Training for Criminal Justice Professionals on Medication-Assisted Treatment. Journal of Addictions & Offender Counseling, 36(1), 13-27.
- [Background] McDowell, I., & Newell, C. (1996). The Short Form 36 Health Survey. Measuring Health, 446-454.
- [Background] McKay, J. R. (2009). Treating substance use disorders with adaptive continuing care. Washington, D.C.: American Psychological Association.
- [Background] McKay JR, Lynch KG, Shepard DS, Morgenstern J, Forman RF, Pettinati HM. Do patient characteristics and initial progress in treatment moderate the effectiveness of telephone-based continuing care for substance use disorders? Addiction. 2005 Feb;100(2):216-26. doi: 10.1111/j.1360-0443.2005.00972.x. PMID 15679751
- [Background] Murphy, S. A., & McKay, J. R. (2004). Adaptive treatment strategies: an emerging approach for improving treatment effectiveness. Clinical Science, 12, 7-13.
- [Background] National Institute on Drug Abuse. (2018). Overdose death rates. Retrieved from https://www.drugabuse.gov/related-topics/trends-statistics/overdose-death-rates.
- [Background] Philadelphia DBHIDS. (2018). Mayor's Task Force to Combat the Opioid Epidemic in Philadelphia. The Opioid Epidemic in Philadelphia. Philadelphia, PA: City of Philadelphia DBHIDS. Mar p. 40.
- [Background] Philadelphia Department of Public Health (2018). Opioid Surveillance. Retrieved from https://hip.phila.gov/datareports/opioid
- [Background] Reid R, Pipe A, Higginson L, Johnson K, D'Angelo MS, Cooke D, Dafoe W. Stepped care approach to smoking cessation in patients hospitalized for coronary artery disease. J Cardiopulm Rehabil. 2003 May-Jun;23(3):176-82. doi: 10.1097/00008483-200305000-00003. PMID 12782900
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] Schwartz RP, Kelly SM, Mitchell SG, Gryczynski J, O'Grady KE, Gandhi D, Olsen Y, Jaffe JH. Patient-centered methadone treatment: a randomized clinical trial. Addiction. 2017 Mar;112(3):454-464. doi: 10.1111/add.13622. Epub 2016 Nov 10. PMID 27661788
- [Background] Seth P, Scholl L, Rudd RA, Bacon S. Overdose Deaths Involving Opioids, Cocaine, and Psychostimulants - United States, 2015-2016. MMWR Morb Mortal Wkly Rep. 2018 Mar 30;67(12):349-358. doi: 10.15585/mmwr.mm6712a1. PMID 29596405
- [Background] Substance Abuse and Mental Health Services Administration. (2011). Consumer-operated services: the evidence (HHS Pub. No. SMA-11-4633). Rockville, MD: U.S. Department of Health and Human Services.
- [Background] Substance Abuse and Mental Health Services Administration. (2015). Medication and counseling treatment. Retrieved from https://www.samhsa.gov/medication-assisted-treatment/treatment.
- [Background] Substance Abuse and Mental Health Services Administration. (2017). Behavioral health treatments and services. Retrieved from https://www.samhsa.gov/treatment
- [Background] Taylor, P. (2014). Drug court practitioner fact sheet: building recovery oriented systems of care for drug court participants. National Drug Court Institute. Retrieved from http://www.ndci.org/sites/default/files/nadcp/Recovery-Oriented%20Systems%20of%20Care.pdf.
- [Background] Marlowe, D. B., & Wong, C. J. (2008). Contingency management in adult criminal drug courts. Contingency management in substance abuse treatment, 334-354.
- [Background] Dugosh, K. D. & Festinger, D. S. (2017). Ohio Addiction Treatment Program final report. Retrieved from http://mha.ohio.gov/Portals/0/assets/Initiatives/ATPP/Final-ATP-Evaluation-Report.pdf
- [Background] Drug Enforcement Administration. (2017). Analysis of overdose deaths in Pennsylvania, 2016 (DEA-PHL-DIR- 034-17). Pittsburgh, PA: University of Pittsburgh.
- [Background] Diggle, P. J., Heagerty, P., Liang, K. Y., & Zeger, S. L. (2002). Analysis of longitudinal data. Oxford, UK: Oxford University Press. Drug Addiction Treatment Act of 2000, H.R. 2634, 106th Cong. (2000).
- [Background] Department of Health and Human Services. (2016). Medication assited treatment for opioid use disorder (42 CFR Part 8, RIN 0930-AA22). Rockville, MD: Substance Abuse and Mental Health Services Administration.
- [Background] Department of Health and Human Services. (2013). Addressing current drug abuse in the United States: current activities and future opportunities. Retrieved from: https://www.cdc.gov/drugoverdose/pdf/hhs_prescription_drug_abuse_report_09.2013.pdf
- [Background] Comprehensive Addiction Recovery Act of 2015, H.R. 953, 114th Cong. (2015). Comprehensive Addiction Recovery Act of 2016, S.524, 114th Cong. (2016).
- [Background] Centers for Disease Control and Prevention. (2018). State of the state of Pennsylvania. Retrieved from https://www.cdc.gov/nchs/pressroom/states/pennsylvania/pennsylvania.htm
- [Background] Centers for Disease Control and Prevention. (2017). Wide-ranging online data for epidemionlogic research (WONDER). Atlanta, GA: CDC, National Center for Health Statistics. Retrieved from http://wonder.cdc.gov.
- [Background] Centers for Disease Control and Prevention (2018). Provisional Drug Overdose Death Counts. Retrieved from https://www.cdc.gov/nchs/nvss/vsrr/drug-overdose-data.htm
- [Background] Blash, L., Chan, K., & Chapman, S. (2015). The peer provider workforce in behavioral health: a landscape analysis. San Francisco, CA: UCSF Health Workforce Research Center on Long-Term Care.
- [Background] American Society of Addiction Medicine. (2013). Advancing access to addiction medications: implications for opioid addiction treatment. Chevy Chase, MD.
- [Background] Allison, P. D. (2010). Survival analysis using SAS: a practical guide, 2nd edition. Cary, NC: SAS Institute, Inc.
- [Derived] Lent MR, Dugosh KL, Hurstak E, Callahan HR, Mazur K; Greater Philadelphia Opioid Use Disorder Research Group. Prevalence and predictors of suicidality among adults initiating office-based buprenorphine. Addict Sci Clin Pract. 2023 Jun 1;18(1):37. doi: 10.1186/s13722-023-00393-y. PMID 37264472
- [Derived] Lent MR, Gaither-Hardy D, Favor KE, Harris D, Cos TA, Millard C, Kone Z, Van Riper A, Dugosh KL. The development, implementation and early learnings of a training program to advance interest in behavioral research careers among undergraduate BIPOC students majoring in psychology. BMC Med Educ. 2023 Mar 15;23(1):160. doi: 10.1186/s12909-023-04104-8. PMID 36922813